CLINICAL TRIAL: NCT03914053
Title: Balancing of Patients Treated by Vitamin K Antagonists (VKAS) in General Medicine : Study ok Variables Influencing the Time Paid in the Therapeutic Target
Brief Title: Balancing of Patients Treated by Vitamin K Antagonists (VKAS) in General Medicine
Acronym: VKA
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL17_0238
Record Dates: First submitted 2019-04-09; First posted 2019-04-12 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2017-07

CONDITIONS: Thromboembolism
MeSH Terms: conditions — Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Despite the rise in prescriptions for direct oral anticoagulants,Vitamin K antagonists(VKA) remains the most prescribed treatment for treating and preventing long-term thromboembolic events. They remain the most important drugs of iatrogenic accidents despite the means deployed by the health authorities. The balance of the patients under VKA can be appreciated thanks to the time spent in the therapeutic zone or TTR which is correlated with the risk of occurrence of haemorrhagic or thrombotic events.

DETAILED DESCRIPTION:
Despite the rise in prescriptions for direct oral anticoagulants, Vitamin K antagonists (VKA) remains the most prescribed treatment for treating and preventing long-term thromboembolic events. They remain the most important drugs of iatrogenic accidents despite the means deployed by the health authorities. The balance of the patients under VKA can be appreciated thanks to the time spent in the therapeutic zone or TTR which is correlated with the risk of occurrence of haemorrhagic or thrombotic events.

The management of VKA in France seems hardly comparable to that of the neighboring countries in front of:

* A TTR estimated at 60%.
* Majority management of anticoagulant treatments by general practitioners.
* The weak development of clinics anticoagulants.
* The takeoff of direct oral anticoagulant prescriptions.
* Preponderance of fluindione prescriptions among the various oral anticoagulants.

It therefore seems interesting to study a cohort of French patients under VKA. Through the calculation of the TTR, the investigators will be able to draw a picture of the balance of the anticoagulant treatment and try to identify factors that can influence it.

ELIGIBILITY:
Inclusion Criteria:

* Patient treated with VKA.
* Realization of INR in one of the labs of the territory of LaboSud Oc biology between 1 September 2015 and 13 January 2016.

Exclusion Criteria:

* Less than 3 INR during the data collection period (TTR calculation not possible).
* Time greater than 56 days between two INRs (calculation of the invalid TTR).
* Interrupted treatment (calculation of invalid TTR).
* Lack of information about the patient

Age Groups: Child, Adult, Older Adult
Study Population: Patient treated with VKA
Sampling Method: Probability Sample
Enrollment: 3387 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
time spent in the therapeutic range (TTR) | 1 day
  calculating their time spent in the therapeutic range (TTR).

CONTACTS AND LOCATIONS:
Overall Officials: Emile Emile, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC